CLINICAL TRIAL: NCT00760227
Title: Testing the Effectiveness of Child and Parent-Targeted Health Promotion Interventions in Pediatric Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: HOBIT3
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Bone Marrow; Stem Cell Transplant
MeSH Terms: interventions — Massage; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: HPI-C (Other): Child Intervention Only Group
  Interventions: Other: Massage Therapy; Other: Humor Therapy
- 2: HPI-CP (Other): Parent and Child Intervention Group
  Interventions: Other: Massage Therapy; Other: Relaxation Therapy
- 3: SC (No Intervention): Standard Care Control Group- No Intervention

INTERVENTIONS:
Other: Massage Therapy — Patient and parents will meet with a licensed massage therapist at the time of admission. During the session, the therapist will introduce them to the rationale of the massage intervention before moving on to provide the initial massage session. Each session will last approximately 1/2 hour. Massage sessions will be scheduled 3x/week from admission through week +3.
  Arms: 1: HPI-C; 2: HPI-CP
Other: Humor Therapy — For this component will will utilize a humor cart, stocked with humorous video shorts, books, gags, props and games.
  Arms: 1: HPI-C
Other: Relaxation Therapy — In the initial session held near the time of admission, parents will meet with the RA therapist, who will describe relaxation response and the benefits of a regular practice of relaxation techniques. They will be led through a modified progressive muscle relaxation induction, using breath awareness and muscle release, followed by guided imagery.
  Arms: 2: HPI-CP

SUMMARY:
The overall aim of the proposed project is to evaluate the impact of a health promotion intervention for children undergoing bone marrow or stem cell transplant (BMT). The intervention is complementary in nature, designed to increase the experience of positive affect and reduce somatic distress and mood disturbance, that is, to improve overall child well-being. The study will utilize a positive psychology model, exploring the hypothesis that improved outcomes will be mediated by the increased experience of positive affect states brought about by the intervention. The primary focus is on a child-targeted intervention that includes massage therapy and humor therapy. The study will also assess whether the addition of a similar parent-targeted intervention involving massage therapy and relaxation training will provide significant benefits beyond those provided by the child-targeted intervention alone. The study will utilize a 3-group design, with participants randomized to receive:1) a child-targeted intervention (HPI-C); 2) a child targeted intervention plus a parent-targeted intervention (HPI-CP); 3) standard care (SC). Primary outcomes include child positive affect, somatic distress and mood disturbance, as well as measures of parental positive affect and distress. Additional objectives of the study include examining the impact of the intervention on short-term medical outcomes, as well as measures of child health-related quality of life and parent and child post-traumatic stress symptoms (PTSS) at 6 months post-BMT. Analyses will explore hypotheses specific to the positive psychology model, testing the role of positive affect and dispositional optimism as mediators and moderators of the intervention on child and parent well-being. We will also obtain pilot data examining the effect of the interventions on neuroendocrine and neuroimmune markers of stress.

DETAILED DESCRIPTION:
Treatment Plan: Interventions involve 3 components, Massage Therapy, Humor Therapy, and Relaxation Therapy, as described below:

Massage Therapy Patient and parents will meet with a licensed massage therapist at the time of admission. During the session, the therapist will introduce them to the rationale of the massage intervention before moving on to provide the initial massage session. Each session will last approximately 1/2 hour. Massage sessions will be scheduled 3x/week from admission through week +3.

Humor Therapy For this component will utilize a humor cart, stocked with humorous video shorts, books, gags, props and games.

Relaxation Therapy In the initial session held near the time of admission, parents will meet with the RA therapist, who will describe relaxation response and the benefits of a regular practice of relaxation techniques. They will be led through a modified progressive muscle relaxation induction, using breath awareness and muscle release, followed by guided imagery.

ELIGIBILITY:
Inclusion Criteria:

For Child Participants:

* Age 6-18 years inclusive.
* Scheduled to undergo allogeneic or autologous stem cell transplant.
* Anticipated hospital stay of at least 3 weeks.
* English speaking

For Resident Parent Participants:

* Parent speaks and reads English.
* Parent will be a primary caregiver for child during BMT.
* Parent will be available for the duration of transplant hospitalization.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To test the effectiveness of the health-promotion interventions in improving patient and parent well-being during the acute phase of BMT. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sean Phipps, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (4):
- United States (3):
  - Columbus Children's Research Institute, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org